CLINICAL TRIAL: NCT05874544
Title: Rifabutin-containing Triple Therapy for Helicobacter Pylori Rescue Treatment: a Randomized Controlled Trial
Brief Title: Rescue Therapy for Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjhy20230001
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; rescue therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Tetracycline; Metronidazole; Amoxicillin; Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tetracycline Bismuth Quadruple Therapy (Active Comparator): Vonoprazan 20mg bid, Bismuth Potassium Citrate 110mg qid, Tetracycline 500mg qid, Metronidazole 400mg qid
  Interventions: Drug: Vonoprazan; Drug: Bismuth Potassium Citrate; Drug: Tetracycline; Drug: Metronidazole
- Rifabutin Triple Therapy (Experimental): Vonoprazan 20mg bid, amoxicillin 1000mg tid, rifabutin 150mg bid
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: Rifabutin
- Dual Therapy (Experimental): Vonoprazan 20mg bid, amoxicillin 1000mg tid
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin

INTERVENTIONS:
Drug: Vonoprazan — Proton pump inhibitor
Drug: Bismuth Potassium Citrate — Gastric mucosal protective drug with anti-H. pylori effect
  Arms: Tetracycline Bismuth Quadruple Therapy
Drug: Tetracycline — Antibiotics for H. pylori eradication
  Arms: Tetracycline Bismuth Quadruple Therapy
Drug: Metronidazole — Antibiotics for H. pylori eradication
  Arms: Tetracycline Bismuth Quadruple Therapy
Drug: Amoxicillin — Antibiotics for H. pylori eradication
  Arms: Dual Therapy; Rifabutin Triple Therapy
Drug: Rifabutin — Antibiotics for H. pylori eradication
  Arms: Rifabutin Triple Therapy

SUMMARY:
Dual therapy containing vonoprazan and amoxicillin had showed excellent eradication results with Helicobacter pylori first-line treatment. However, no study has examined its efficacy for H. pylori rescue treatment. Rifabutin has low antibiotic resistance, superior antibacterial activity in vitro, and stability in the gastric acid environment. Several studies have confirmed the efficacy of rifabutin-containing triple therapy as a first-line or rescue treatment for H. pylori. The purpose of this study was to evaluate the efficacy and safety of dual therapy vesus rifabutin-containing triple therapy versus classical bismuth-containing quadruple therapy as rescue therapy for the eradication of refractory Helicobacter pylori.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to participate in the study and to sign and give informed consent
* Confirmed H. pylori infection and with previous treatment experience

Exclusion Criteria:

* subjects naive to H. pylori treatment,
* under 18 or over 80 years old
* history of gastrectomy
* pregnant or lactating women
* Previous history of tuberculosis
* Allergy to any of the study drugs
* severe systemic diseases or malignancy
* administration of antibiotics, bismuth, antisecretory drugs, or Chinese herb medicine in the preceding 8 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | Within 7 days after completion of therapy
  The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or severe" (causing considerable interference with daily activities). In addition, blood test were messured to access function of liver and kidney.
Compliance rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Songjiang District Central Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Zhejiang University school of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No